CLINICAL TRIAL: NCT02101229
Title: Diabeloop WP6-1 : Validation of the Artificial Pancreas Diabeloop Algorithm in the Hospital
Brief Title: Validation of the Artificial Pancreas Diabeloop Algorithm in the Hospital
Acronym: WP6-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013-A01657-38
Record Dates: First submitted 2014-03-21; First posted 2014-04-02 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes
Keywords: Glycemic control algorithm; closed loop; artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- unsual treatment (No Intervention): The patient will have his usual treatment in this arm
- The Diabeloop algorithm (Experimental): In this arm, the insulin Asp(B28) dose is calculated by the algorithm based on the usual treatment of the patient, the ratio I / C, the intensity of physical activity and blood glucose sensor.
  Interventions: Drug: Insulin, Asp(B28)-

INTERVENTIONS:
Drug: Insulin, Asp(B28)- — the insulin dose is calculated by the "Diabeloop" algorithm and then administered to the patient
  Other Names: NovoRapid insulin
  Arms: The Diabeloop algorithm

SUMMARY:
To assess whether the DIABELOOP algorithm provides better glycemic control than the usual algorithm of T1D patients on pump therapy:

* at meals, with CHO roughly assessed by the patient.
* during and after physical activity sessions qualified as moderate by the patient.

Primary endpoint : time within the glycemic reference range. The study will be conduct with 15 patients at the following investigation centers : Corbeil Hospital, CHU of Grenoble, and CHU of Montpellier.

DETAILED DESCRIPTION:
The 15 patients will have 2 visits during 24 hours (day and night), once with their usual algorithm and once with the Diabeloop system.

ELIGIBILITY:
Inclusion Criteria:

* Patient type 1 diabetic for at least one year
* Patient treated by external insulin pump for at least 6 months
* Patients with HbA1c <9%
* Patient affiliated with Social Security.
* Patient able to perform two tests of physical activity of 30 minutes (one event in each treatment period);
* aged at least 18 years Patient;
* Patient who signed consent

Exclusion Criteria:

* All serious disease that could interfere with the study
* BMI > 30 kg/m2
* insulin requirement > 2 U/kg/day
* Patient benefiting from a measure of legal protection;
* Pregnant or likely to be women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Time spent in blood glucose range [70-180 mg/dl] | up to 24 hours after each treatment period
  comparing the time spent in [70-180 mg/dl] with usual algorithm vs Diabeloop algorithm.

SECONDARY OUTCOMES:
Time spent Blood Glucose range [80-140 mg/dl] | 24 hours after each treatment period
  Comparing the time spent in range [80-140 mg/dl] with usual algorithm vs Diabeloop algorithm
time spent below 70 mg/dl and above 180 mg/dl | up to 24 hours after each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia FRANC, MD, Principal Investigator — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète; Ahmed DAOUDI, MD, Principal Investigator — Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète; Pierre-Yves BENHAMOU, Pr, Principal Investigator — CHU of Grenoble; Sandrine LABLANCHE, MD, Principal Investigator — CHU of Grenoble; Eric RENARD, Pr, Principal Investigator — CHU of Montpellier; Anne FARRET, MD, Principal Investigator — CHU of Montpellier
Locations (3):
- France (3):
  - Centre Hospitalier du Sud Francillien, Évry
  - University Hospital of Grenoble, Grenoble
  - University Hospital of Montpellier, Montpellier